CLINICAL TRIAL: NCT03410914
Title: A Single-arm Phase II Trial of Intra-operative Application of HEMOPATCH to the Pancreatic Stump to Prevent Post-operative Pancreatic Fistula Following Distal Pancreatectomy
Brief Title: Intra-operative Application of HEMOPATCH to the Pancreatic Stump to Prevent Post-operative Pancreatic Fistula Following Distal Pancreatectomy
Acronym: PATCH-DP
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sunnybrook Health Sciences Centre (Other)
Collaborators: Baxter Healthcare Corporation (Industry); Hamilton Health Sciences Corporation (Other); The Ottawa Hospital (Other); Kingston Health Sciences Centre (Other); Royal University Hospital Foundation (Other); London Health Sciences Centre (Other); University Health Network, Toronto (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 346-2017
Record Dates: First submitted 2018-01-19; First posted 2018-01-25 (Actual); Results first posted 2021-08-09 (Actual); Last update posted 2021-11-03 (Actual); Status verified 2021-10

CONDITIONS: Pancreas Cancer; Pancreas Disease; Pancreas Adenocarcinoma; Pancreas; Fistula; Surgery; Surgery--Complications; Surgery Site Fistula
Keywords: Hemopatch
MeSH Terms: conditions — Pancreatic Neoplasms; Pancreatic Diseases; Pancreatic Fistula

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Hemopatch (Experimental): Application of hemopatch to the divided end of the pancreas during surgery
  Interventions: Device: Hemopatch

INTERVENTIONS:
Device: Hemopatch — Application of hemopatch to the divided end of the pancreas during surgery.

SUMMARY:
Despite improvements and advances in pancreas surgery, about 30-35% of patients who have pancreas surgery develop a type of complication called a pancreatic fistula. A pancreatic fistula occurs when fluid produced by the pancreas leaks into the abdomen after pancreas surgery. Patients who develop a pancreatic fistula can have poor short-term and long-term consequences.We are studying the effect of a medical device named HEMOPATCH on the development and seriousness of pancreatic fistulas. HEMOPATCH is a thin, flexible bovine protein-based pad that may improve tissue sealing where it is applied during surgery. Some small studies called case studies of between 2 and 7 patients, and two clinical trials have shown that HEMOPATCH is effective at stopping bleeding and reducing drain output after some types of surgery. However, there have been no completed clinical trials using HEMOPATCH to prevent or reduce pancreatic fistulas in patients having pancreas surgery, so we don't know if it works in this setting. Health Canada has approved the use of HEMOPATCH as a device to stop bleeding or seal other bodily fluids for procedures in which the control of bleeding or leakage of other body fluids or air by standard surgical techniques are either ineffective or impractical.

ELIGIBILITY:
Inclusion Criteria:

* Scheduled to undergo distal pancreatectomy surgery that is open or laparoscopic, with or without splenectomy
* Age ≥ 18 years
* Able and willing to comply with study procedures and follow-up examinations contained within the written consent form

Exclusion Criteria:

* Contraindication to placement of HEMOPATCH tissue sealant including: 1) Known hypersensitivity to bovine proteins; 2) Known hypersensitivity to brilliant blue [FD&C Blue No.1 (Blue 1)]; 3) Presence of an active infection; and 4) Known pregnancy or lactation (a negative urine pregnancy test must be obtained for women of child bearing potential during the pretreatment evaluation)
* Participating in another interventional trial that may result in co-intervention or contamination (to be determined by sponsor)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2018-08-13 (Actual); Primary Completion 2020-10-03 (Actual); Study Completion 2020-10-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paul Karanicolas, MD, Principal Investigator — Sunnybrook Health Sciences Centre
Locations (7):
- Canada (7):
  - Hamilton Health Sciences, Hamilton, Ontario
  - Kingston General Hospital, Kingston, Ontario
  - London Health Sciences Centre, London, Ontario
  - The Ottawa Hospital, Ottawa, Ontario
  - University Health Network, Toronto, Ontario
  - Sunnybrook Health Sciences Centre, Toronto, Ontario
  - Royal University Hospital, Saskatoon, Saskatchewan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bubis LD, Behman R, Roke R, Serrano PE, Khalil JA, Coburn NG, Law CH, Bertens K, Martel G, Hallet J, Marcaccio M, Balaa F, Quan D, Gallinger S, Nanji S, Leslie K, Tandan V, Luo Y, Beck G, Skaro A, Dath D, Moser M, Karanicolas PJ; HPB CONCEPT team. PATCH-DP: a single-arm phase II trial of intra-operative application of HEMOPATCH to the pancreatic stump to prevent post-operative pancreatic fistula following distal pancreatectomy. HPB (Oxford). 2022 Jan;24(1):72-78. doi: 10.1016/j.hpb.2021.05.007. Epub 2021 Jun 9. PMID 34176743

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 78 patients were assessed for eligibility at 7 hepatopancreaticobiliary centres in Canada. Of these, 52 patients met the inclusion criteria and consented to trial participation. These 52 participants were enrolled and allocated to the investigational Hemopatch intervention.
Period: Overall Study
Arm/Group | Hemopatch
Started | 52
Completed | 52
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Hemopatch
Number analyzed (Participants) | 52
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 69 [59 to 74]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20
  Male | 32
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Canada | 52

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With a Clinically Significant Post-operative Pancreatic Fistula (POPF)
Description: Incidence of clinically-significant POPF - defined as ISGPS Grade B or C POPF. Determination of Grade B or C POPF was made on the basis of confirmation of presence of pancreatic fistula (any measurable volume of drain fluid on or after postoperative day 3, with an amylase content greater than 3 times the upper normal serum value) in conjunction with a review of participants' postoperative clinical course.
Time Frame: Within 90 days post-operatively
Measure: Count of Participants; unit: Participants
Arm/Group | Hemopatch
Number analyzed (Participants) | 52
Participants | 13

2. Secondary Outcome: Number of Participants With a Post-operative Pancreatic Fistula (POPF)
Description: Incidence of any POPF - defined as International Study Group Pancreatic Fistula (ISGPF) all grades (A, B, C). Determination of POPF grade was made on the basis of confirmation of presence of pancreatic fistula (any measurable volume of drain fluid on or after postoperative day 3, with an amylase content greater than 3 times the upper normal serum value) in conjunction with a review of participants' postoperative clinical course.
Time Frame: Within 90 days post-operatively
Measure: Count of Participants; unit: Participants
Arm/Group | Hemopatch
Number analyzed (Participants) | 52
Participants | 25

3. Secondary Outcome: Number of Participants Who Experienced Post-Operative Complications
Description: Postoperative complications graded using the Clavien-Dindo system - participants experiencing a Clavien-Dindo complication of greater than or equal to 3 were counted (grade 3 or higher is typically indicated by a procedural intervention to treat the post-operative complication). This grading system was used as a measure of 90-day postoperative morbidity.
Time Frame: Within 90 days post-operatively
Measure: Count of Participants; unit: Participants
Arm/Group | Hemopatch
Number analyzed (Participants) | 52
Participants | 14

4. Secondary Outcome: 90-Day Mortality Count
Description: Indicated by death within 90-days after surgery.
Time Frame: Within 90 days post-operatively
Measure: Count of Participants; unit: Participants
Arm/Group | Hemopatch
Number analyzed (Participants) | 52
Participants | 2

5. Secondary Outcome: Average Length of Stay in Hospital
Description: Number of days from date of surgery (POD0) to the date of discharge
Time Frame: Within 90 days post-operatively
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Hemopatch
Number analyzed (Participants) | 52
days | 6 [4 to 8]

ADVERSE EVENTS:
Time Frame: Adverse events were recorded up until 90 days post-operative.
Arm/Group | Hemopatch
All-Cause Mortality (participants affected / at risk) | 2/52
Serious Adverse Events (participants affected / at risk) | 14/52
Other Adverse Events (participants affected / at risk) | 21/52
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Hemopatch (N=52)
Atrial Fibrillation (Cardiac disorders) | 1 (1)
Grade B POPF (Hepatobiliary disorders) | 6 (6)
Grade C POPF (Hepatobiliary disorders) | 1 (1)
Intra-Abdominal Abscess (Infections and infestations) | 1 (1)
Respiratory Distress (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Bleed (General disorders) | 3 (3)
Colonic Anastomotic Leak (Gastrointestinal disorders) | 2 (2)
Pancreatitis (Hepatobiliary disorders) | 1 (1)
Bile Leak (Hepatobiliary disorders) | 1 (1)
Disseminated Intravascular Coagulation (Blood and lymphatic system disorders) | 1 (1)
Urinary Retention (Renal and urinary disorders) | 1 (1)
Acute Coronary Syndrome/NSTEMI (Cardiac disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Hemopatch (N=52)
Deep Wound Infection (Infections and infestations) | 3 (3)
Grade B POPF (Hepatobiliary disorders) | 6 (6)
Biochemical Leak (Grade A POPF) (Hepatobiliary disorders) | 12 (12)
Neurological (Psychiatric disorders) | 4 (4)
Ileus (Gastrointestinal disorders) | 3 (3)

LIMITATIONS AND CAVEATS:
Broad inclusion criteria does not permit specific evaluation of patient subgroups given overall small sample size. Small sample size also introduces the potential for oversampling of high-risk cases, such as those requiring multivisceral resection.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-04-18): https://cdn.clinicaltrials.gov/large-docs/14/NCT03410914/Prot_SAP_000.pdf